CLINICAL TRIAL: NCT07383688
Title: Survey Study of Subjects Receiving Replacement of Traditional Sacral Neuromodulation (SNM) With the Neuspera SNM System
Brief Title: Neuspera Replacement Survey Study
Status: Not yet recruiting | Type: Observational
Sponsor: Neuspera Medical, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: Neuspera Medical (NSM-007)
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Urinary Urge Incontinence
MeSH Terms: conditions — Urinary Incontinence, Urge

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Neuspera Replacement Cohort: Subjects with previous traditional SNM system and now undergoing implant of the Neuspera SNM System
  Interventions: Device: Neuspera Implantable Sacral Neuromodulation System

INTERVENTIONS:
Device: Neuspera Implantable Sacral Neuromodulation System — Stimulation of the Sacral Nerve

SUMMARY:
Single-arm study where subjects' responses to a questionnaire for the traditional Sacral Neuromodulation (SNM) devices will be compared to the responses regarding the Neuspera SNM System.

DETAILED DESCRIPTION:
Subjects will be enrolled in a single-arm study and followed for 1-month after implant of the Neuspera SNM System.

Subjects will complete a questionnaire regarding their experience with the traditional SNM system prior to the Neuspera implant, then undergo an implant of the Neuspera SNM system using standard of care according to the device's commercial labeling.

Up to 20 subjects will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Currently have a traditional SNM device and has decided to have the device replaced with the Neuspera SNM System OR previously had an existing traditional SNM implant that was completely removed within the last year
2. Is 22 years of age or older
3. Had documented at least 50% improvement in UUI episodes on a bladder diary with either a stimulation trial or with their traditional system
4. Is a good surgical candidate and qualified to receive the Neuspera SNM System per the device labeling
5. Is capable of participating in all testing and follow-up clinic visits associated with this clinical study.

Exclusion Criteria:

1. Has a contraindication for the Neuspera SNM System per the device labeling.
2. Has plans to enroll or is currently enrolled in another investigational device or drug trial during his/her participation in this study

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population with 22 years of age or older and who have or have previously had a traditional SNM system.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Primary Study measure | 1 month
  The changes to subject questionnaire responses for the Neuspera SNM system compared to responses regarding traditional SNM systems

CONTACTS AND LOCATIONS:
Overall Officials: Kellen Choi, DO, Principal Investigator — University of Louisville Health System

REFERENCES:
- See also: Neuspera Medical web page — http://neuspera.com